CLINICAL TRIAL: NCT05436470
Title: Treatment (Compassionate) Use of Device - PK Papyrus
Status: Temporarily not available | Type: Expanded Access
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert Starke, Associate Professor, University of Miami
Other Study IDs: 20220552
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pseudoaneurysm, Carotid; Pseudoaneurysm
MeSH Terms: conditions — Carotid Artery Injuries; Aneurysm, False

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Device: PK Papyrus — The PK Papyrus is a balloon mounted stent that will be administered during standard of care treatment of pseudoaneurysms.

SUMMARY:
The purpose of this study is to evaluate the clinical use of the PK Papyrus Coronary Stent Graft System, a Humanitarian Use Device (HUD) approved by the FDA under a Humanitarian Device Exemption.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with traumatic, dissecting, pseudo, or other wide based aneurysms in non-perforator territories or fistulas of the extracranial or intracranial segments of the internal carotid or vertebral artery.

Exclusion Criteria:

1. Patients from special populations including individuals who are not yet adults (infants, children, teenagers).
2. Adults who are cognitively impaired, pregnant women, and prisoners.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Starke, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States